CLINICAL TRIAL: NCT00954122
Title: A 3 Weeks Open Label Study to Evaluate the Efficacy in Agitation and Safety of Quetiapine Fumarate XR in Treatment of Patients With Acute Schizophrenia
Brief Title: Efficacy and Safety of SEROQUEL Extended Release (XR) in Acute Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00074
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Acute schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine XR (Experimental): Quetiapine XR 300 mg on day 1, 600 mg on day 2, and 400-800 mg (at investigator's discretion) on day 3 and onwards.
  Interventions: Drug: Quetiapine XR (Seroquel XR)

INTERVENTIONS:
Drug: Quetiapine XR (Seroquel XR) — Tablet, oral, once daily
  Other Names: Seroquel XR

SUMMARY:
The purpose of the study is to determine whether treatment with quetiapine XR (Seroquel XR) tablets for 3 weeks will improve their agitation when they have acute psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Requirement for treatment of acute episode of schizophrenia (according to DSM-IV diagnostic criteria)
* PANSS total score of ³ 75
* CGI > 4

Exclusion Criteria:

* Any DSM-IV (Diagnostic and Statistical Manual of Mental Disorders 4th Edition) Axis I disorder not defined in the inclusion criteria
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Substance or alcohol dependence at enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Hatim Sulaiman,, M Psyc, Principal Investigator — University of Malaya; Badiah Yahya, MD, Principal Investigator — Hospital Permai
Locations (2):
- Malaysia (2):
  - Research Site, Johor Bahru, Johor Bahru
  - Research Site, Kuala Lumpur

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 Years to 65 Years Male & Female Acte schizophrenia (DSM-IV) Positive and Negative Syndrome Scale (PANSS) score at least 75, Clinical Global Impression (CGI)
Pre-assignment Details: 40 patients enrolled, 35 patients randomised and 28 patients completed the study
Groups:
- Quetiapine Fumarate XR: This is a one arm Study. Patients were on quetiapine XR 300 mg on day 1, 600 mg on day 2, and 400-800 mg (at investigator's discretion) on day 3 and onwards
Period: Overall Study
Arm/Group | Quetiapine Fumarate XR
Started | 35
Completed | 28
Not Completed | 7
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 1
Not completed — Safety Reason | 1

BASELINE CHARACTERISTICS:
Arm/Group | Quetiapine Fumarate XR
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.3 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Region of Enrollment [Number; unit: participants]
  Malaysia | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale Excited Component (PANSS-EC) Score
Description: PANSS- Excited Component (EC) subscale score will be calculated by adding together the following item scores: excitement (positive subscale item 4); hostility (positive subscale item 7); tension (general subscale item 4); uncooperativeness (general subscale item 8); poor impulse control (general subscale item 14). This is rated on a 7-point Likert scale from 'absent' to 'extremely severe' (score range 5 to 35 points; mean scores = 20 points clinically corresponds to severe agitation). Lower value gives the better outcome.
Time Frame: Baseline and Day 21
Population: ITT population, which comprise of patients who have baseline and at least ONE (1) set of post-baseline PANSS assessments. No imputation on PANSS-EC score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Quetiapine Fumarate XR: Patients were on quetiapine XR 300 mg on day 1, 600 mg on day 2, and 400-800 mg (at investigator's discretion) on day 3 and onwards
Arm/Group | Quetiapine Fumarate XR
Number analyzed (Participants) | 35
Scores on a scale | -7.5 (4)

2. Secondary Outcome: Change From Baseline to Final Visit at Day 21 in PANSS Positive, General Psychopathological Scores.
Description: Positive scale includes 7 Items (Delusions, Conceptual disorganization, Hallucinations, Hyperactivity, Grandiosity, Suspiciousness/persecution, Hostility)and is calculated by adding the positive subscale item scores. Minimum score is 7, maximum score is 49. General Psychopathology scale:16 items (Somatic concern, Anxiety, Guilt feelings, Tension, Mannerisms and posturing, Depression, Motor retardation, Uncooperativeness, Unusual thought content, Disorientation, Poor attention, Lack of judgment and insight, Disturbance of volition, Poor impulse control, Preoccupation, Active social avoidance). Minimum score is 16, maximum score is 112. The higher score- the worse outcome. The biggest reduction of score from baseline- a better efficacy.
  Measure includes PANSS-Positive (range 8-30), PANSS-General Psychopathological (PANSS-G)(range 17-70), total PANSS score (range 37-143), PANSS aggression, hostility and depression cluster scores (range 4-19).
Time Frame: Baseline and Day 21
Population: ITT population, which comprise of patients who have baseline and at least ONE (1) set of post-baseline PANSS assessments. No imputation on PANSS Negative score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine Fumarate XR
Number analyzed (Participants) | 35
Scores on a scale | -9.3 (5.5)

3. Secondary Outcome: Change From Baseline to Final Visit at Day 21 in PANSS Negative, General Psychopathological Scores
Description: Negative scale includes 7 items (Blunted affect, Emotional withdrawal, Poor rapport, Passive/apathetic social withdrawal, Difficulty in abstract thinking, Lack of spontaneity and flow of conversation, Stereotyped thinking)and is calculated by adding the negative subscale item scores. Minimum score is 7, maximum score is 49. General Psychopathology scale includes 16 Items (Somatic concern, Anxiety, Guilt feelings, Tension, Mannerisms and posturing, Depression, Motor retardation, Uncooperativeness, Unusual thought content, Disorientation, Poor attention, Lack of judgment and insight, Disturbance of volition, Poor impulse control, Preoccupation, Active social avoidance). Minimum score is 16, maximum score is 112. The higher score- the worse outcome. Measure includes PANSS-Negative (range 8-37), PANSS-General Psychopathological (PANSS-G)(range 17-70), total PANSS score (range 37-143), PANSS aggression, hostility and depression cluster scores (range 4-19).
Time Frame: Baseline and Day 21
Population: ITT population, which comprise of patients who have baseline and at least ONE (1) set of post-baseline PANSS assessments. No imputation on PANSS Positive score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine Fumarate XR
Number analyzed (Participants) | 35
Scores on a scale | -5.7 (4.9)

4. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: Positive and Negative Syndrome Scale (PANSS) total score is a medical scale used for measuring symptom severity of patients with schizophrenia. It is calculated by adding together PANSS-Positive (minimum score = 7, maximum score = 49, PANSS-Negative (minimum score = 7, maximum score = 49), PANSS-General Psychopathological (PANSS-G) subscale scores (minimum score = 16, maximum score = 112), supplementary subscale item scores. The minimum is 30, maximum is 210. Total PANSS score classification: Mildly ill 58- 74, Moderately ill 75-94, Markly ill 95- 115, Severely ill >116.
Time Frame: Baseline and Day 21
Population: ITT population, which comprise of patients who have baseline and at least ONE (1) set of post-baseline PANSS assessments. No imputation on PANSS Total score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine Fumarate XR
Number analyzed (Participants) | 35
Scores on a scale | -33.2 (21.3)

5. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity Scale (CGI-S)
Description: Clinical Global Impression, Severity (CGI-S) is a single-item (7-point) scale that evaluates the overall severity of the subject's mental illness. A reduction in score indicates an improvement in the subject's condition. The CGI-S assessment should be based upon the subject's symptoms during the previous week.
  Change from baseline in CGI-S score is calculated by subtracting the CGI-S score at baseline from the CGI-S score at the relevant time point.
Time Frame: Baseline and Day 21
Population: ITT population, which comprise of patients who have baseline and at least ONE (1) set of post-baseline PANSS (Positive and Negative Syndrome Scale) assessments. No imputation on CGI-S score.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine Fumarate XR
Number analyzed (Participants) | 35
scores on a scale | -1.2 (0.9)

6. Secondary Outcome: Change From Baseline in Absolute Clinical Global Impression-Improvement (CGI-I) Scale
Description: Clinical Global Impression, Improvement (CGI-I) is a single-item (7-point) scale that evaluates the overall improvement in the subject's mental. A reduction in score indicates an improvement in the subject's condition. This assessment is based on the improvement since initiation of the study treatment.
  Change in CGI-I score is analyzed by comparing CSI-score at the relevant time point to the baseline CGI-I score.
Time Frame: Baseline and Day 21
Population: ITT population, which comprise of patients who have baseline and at least ONE (1) set of post-baseline PANSS (Positive and Negative Syndrome Scale) assessments. No imputation on CGI-I score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine Fumarate XR
Number analyzed (Participants) | 35
Scores on a scale
  Baseline | 3.9 (0.4)
  Day 21 | 2.4 (1.2)

7. Secondary Outcome: Change of the Positive and Negative Syndrome Scale Excited Component (PANSS-EC) Score Compared From Baseline to Day 21.
Description: Excited Component was used to evaluate the control of agitation and aggression in patients with schizophrenia.
  Difference in mean score at baseline and day 21 is used to assess the improvement. It is shown by reduction in mean score and confirmed by p value lower than 0,05.
  Positive and Negative Syndrome Scale Excited Component (PANSS-EC) is a subscale score which is calculated by adding together the following item scores: excitement (positive subscale item 4); hostility (positive subscale item 7); tension (general subscale item 4); uncooperativeness (general subscale item 8); poor impulse control (general subscale item 14).
  This is rated on a 7-point Likert scale from 'absent' to 'extremely severe' (score range 5 to 35 points; mean scores = 20 points clinically corresponds to severe agitation).
Time Frame: Baseline and Day 21
Population: ITT population, which comprise of patients who have baseline and at least ONE (1) set of post-baseline PANSS assessments. No imputation on Outcome Measurement.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine Fumarate XR
Number analyzed (Participants) | 35
Scores on a scale | -33.2 (21.3)

ADVERSE EVENTS:
Arm/Group | Quetiapine Fumarate XR
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine Fumarate XR (N=35)
Hospitalization (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other